CLINICAL TRIAL: NCT06458985
Title: Disclosure Intervention to Reduce Social Isolation and Facilitate Recovery Among People in Treatment for Opioid Use Disorder
Brief Title: Disclosure Intervention for People in Treatment for Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Brandywine Counseling and Community Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDISCLOSE RCT; R01DA059557 (NIH)
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder
Keywords: disclosure; social isolation; stigma; social support
MeSH Terms: conditions — Opioid-Related Disorders; Social Isolation; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disclosing Recovery (Experimental): Participants complete a one-hour disclosure intervention for people in treatment for opioid use disorder. The intervention is facilitated by a workbook and accompanying worksheet.
  Interventions: Behavioral: Disclosing Recovery: A Decision Aid and Toolkit
- Waitlist Comparator (No Intervention): Participants do not complete the disclosure intervention at their baseline appointment. They are given the opportunity to complete the disclosure intervention at their final appointment.

INTERVENTIONS:
Behavioral: Disclosing Recovery: A Decision Aid and Toolkit — The Disclosing Recovery intervention is designed to help people in treatment for opioid use disorder (1) make key decisions regarding disclosure, including whether, why, what, how, and when to disclose, and (2) build skills to disclose, including planning what to say, practicing disclosure, and preparing for negative responses.
  Other Names: Disclosing Recovery
  Arms: Disclosing Recovery

SUMMARY:
The goal of this clinical trial is to test a disclosure intervention among people in treatment for opioid use disorder. The main question it aims to answer is whether people who receive a disclosure intervention have better treatment- and recovery-related outcomes one year after receiving the intervention. Participants will complete a brief disclosure intervention designed to help them (1) make key disclosures related to disclosure and (2) build skills to disclose. Researchers will compare results to participants in a waitlist comparator condition, who receive the intervention at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Client of Brandywine Counseling & Community Services
* Receiving opioid use disorder treatment at Brandywine Counseling & Community Services
* Considering disclosing one's opioid use disorder history and/or treatment to someone new

Exclusion Criteria:

* Diagnosis of schizophrenia
* Participation in pilot study of intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Retention in treatment | 1 year
  Whether participants are retained in treatment 1 year after baseline
Illicit opioid use | 1 year
  Percentages of drug screens that are positive for illicit opioid use

SECONDARY OUTCOMES:
Recovery capital score | 1 year
  Average scores on recovery capital measure (titled: Brief Assessment of Recovery Capital); items are measured on a 1-5 point Likert-type scale, and composite scores range from 1-5. Higher values indicate greater recovery capital.
Quality of life score | 1 year
  Average scores on quality of life measure (titled: European Health Interview Survey-Quality of Life - 8 item); items are measured on a 1-5 point Likert-type scale, and composite scores range from 1-5. Higher scores indicate greater quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Brandywine Counseling & Community Services, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this project will be shared via the National Addiction & HIV Data Archive Program (NAHDAP), which is hosted by the Inter-university Consortium for Political and Social Research (ICPSR). Responses to surveys and medical record data will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available no later than when the primary outcome paper is published or when the award ends, whichever comes first. The data will be shared indefinitely.
Access Criteria: Data will be accessible through the National Addiction & HIV Data Archive Program (NAHDAP). NAHDAP will make data available via restricted-use files (which will require a signed Restricted Data Use Agreement between the requestor's institution and the University of Michigan as well as an application to request access). ICPSR/NAHDAP will approve or deny access based on the results of the application review.